CLINICAL TRIAL: NCT00241215
Title: Probe Study to Evaluate the Efficacy of Botulinum Toxin Serotype A Injections for Cervicobrachial Myofascial Syndrome
Brief Title: Study to Evaluate the Efficacy of Botulinum Toxin Serotype A Injections for Cervicobrachial Myofascial Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, F. Michael Ferrante, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: UCLA#03-03-061-03A
Record Dates: First submitted 2005-10-17; First posted 2005-10-18 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Cervicobrachial Neuralgia; Myofascial Pain Syndromes
Keywords: Botulinum toxin serotype A; Cervicobrachial syndrome; Myofascial pain; Cervicothoracic myofascial pain; Propulsion; Postural abnormality
MeSH Terms: conditions — Brachial Plexus Neuritis; Myofascial Pain Syndromes

INTERVENTIONS:
Drug: Botulinum toxin serotype A

SUMMARY:
Several studies have previously examined the use of botulinum toxin serotype A for myofascial pain of the neck and shoulders (cervicobrachial syndrome). These studies have suffered from:

1. inclusion of confounding conditions in the proband group, and
2. inability to identify predictors of response.

This study attempts to define the characteristics of responders to botulinum serotype A for myofascial pain of the neck and shoulders (cervicobrachial syndrome).

DETAILED DESCRIPTION:
Design: Single-center, double-blind, placebo-controlled, enriched trial.

Subjects will wash-out of their existing pain medications at least 2 weeks prior to baseline visit. At baseline, patients with a Numerical Pain Rating of 4 or greater will be injected with Botulinum Toxin Serotype A. At 14 weeks postinjection, those who at the 6 weeks post-injection visit had at least a 50% decrease in their pain outcome measures will be randomized into one of two treatment groups. Group 1 will receive a second BTX injection while group 2 will receive an injection of saline and both groups will be followed for an additional 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-65 years.
2. Patients present with bilateral posterior neck/cervical muscle pain for greater than 8 weeks
3. Patients have numerical pain rating of 4 or greater
4. Patients willing to adhere to a physical therapy program of 2-3 visits for myofascial release and also home stretching exercises for the length of the study
5. Subjects willing to discontinue all pain medications except ibuprofen and a non-opioid rescue medication for the duration of the study.
6. Women of child-bearing potential must be using a reliable means of contraception and have a negative urine pregnancy test prior to injection of BOTOX.

Exclusion Criteria:

1. Subjects currently taking schedule II narcotics
2. No new non-pain medications or change in non-pain medications within 2 months of screening or throughout the study
3. Pregnant or breastfeeding women
4. Use of investigational drugs within one month of study
5. Involvement in litigation surrounding neck pain
6. Significant medical or psychiatric disease
7. Patients with clinical depression (Beck's Depression score)
8. Alcohol or drug abuse, in the opinion of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2003-06; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Numerical pain rating
Brief Pain Inventory
Neck Disability Index
Cervical range of motion
Number of trigger points
Postural exam

SECONDARY OUTCOMES:
Pain Diary and medications use
Short Form (SF)-36

CONTACTS AND LOCATIONS:
Overall Officials: F. Michael Ferrante, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Pain Management Center, Santa Monica, California, United States

REFERENCES:
- [Result] Ferrante FM, Bearn L, Rothrock R, King L. Evidence against trigger point injection technique for the treatment of cervicothoracic myofascial pain with botulinum toxin type A. Anesthesiology. 2005 Aug;103(2):377-83. doi: 10.1097/00000542-200508000-00021. PMID 16052120